CLINICAL TRIAL: NCT01580293
Title: A Phase II/III, Multicenter, Partially Randomized, Open Label Trial Investigating Safety and Efficacy of On-demand and Prophylactic Treatment With BAY94-9027 in Severe Hemophilia A
Brief Title: A Trial Investigating Safety and Efficacy of Treatment With BAY94-9027 in Severe Hemophilia A
Acronym: PROTECT-VIII
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13024; 2011-005210-11 (EudraCT Number)
Record Dates: First submitted 2012-03-28; First posted 2012-04-19 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hemophilia A
Keywords: Hemophilia A, factor VIII, prophylaxis
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): On-demand treatment of BAY94-9027 at individual dose and number of infusions based upon location and severity of bleeds
  Interventions: Biological: BAY94-9027
- Arm 2 (Experimental): Prophylaxis treatment of BAY94-9027; 2 infusions per week over 10 weeks followed by 2 infusions per week over 26 weeks in the main trial; and at least 1 day per week in the extension for at least 100 ED
  Interventions: Biological: BAY94-9027
- Arm 3 (Experimental): Prophylaxis treatment of BAY94-9027; 2 infusions per week over 10 weeks followed by infusion every 5 days over 26 weeks in the main trial; and at least 1 day per week in the extension for at least 100 ED
  Interventions: Biological: BAY94-9027
- Arm 4 (Experimental): Prophylaxis treatment of BAY94-9027; 2 infusions per week over 10 weeks followed by infusion every 7 days over 26 weeks in the main trial; and at least 1 day per week in the extension for at least 100 ED
  Interventions: Biological: BAY94-9027

INTERVENTIONS:
Biological: BAY94-9027 — Intravenous infusion of BAY94-9027

SUMMARY:
Haemophilia A is an inherited disorder in which one of the proteins, Factor VIII, needed to form blood clots is missing or not present in sufficient levels. In a person with haemophilia A, the clotting process is slowed and the person experiences bleeds that can result in serious problems and potential disability.

The current standard treatment for severe haemophilia A is regularly scheduled infusion of FVIII to keep levels high enough to prevent bleeding. Due to the short half-life of FVIII, prophylaxis may require treatment as often as every other day.

In this trial safety and efficacy of a long-acting recombinant factor VIII molecule is evaluated in subjects with severe Hemophilia A.

120-140 patients will receive open label treatment with long-acting rFVIII either on-demand to treat bleeds or prophylactically for 36 weeks in the main trial plus an optional extension to continue treatment for at least 100 total exposure days (ED). Patients on prophylactic treatment will receive study drug at dosing intervals between once and twice a week depending on their observed bleeding. Patients will attend the treatment centre for routine blood samples and be required to keep an electronic diary.

Male patients aged 12-65, with severe hemophilia A, previously treated with FVIII for at least 50 exposure days may be eligible for this study.

DETAILED DESCRIPTION:
Subjects in prophylactic treatment arms will undergo clinical evaluation at 10 weeks. Those with adequate control of bleeding will undergo randomization to every 5 or 7 day infusion. Those with continued bleeding will remain in treatment arm and have an increase in dose.

Part B-major surgery - optional sub study included to collect information on efficacy of BAY94-9027 in major surgical setting. Due to rarity of surgery in this population, enrollment to this sub-study may be independent of participation in main study.

ELIGIBILITY:
Inclusion Criteria:

* Male; 12-65 years of age
* Subjects with severe hemophilia A
* Previously treated with factor VIII for a minimum of 150 exposure days

Exclusion Criteria:

* Inhibitors to FVIII (current evidence or history)
* Any other inherited or acquired bleeding disorder in addition to Hemophilia A
* Platelet count < 100,000/mm3
* Creatinine > 2x upper limit of normal or AST/ALT (aspartate aminotransferase/alanine aminotransferase) > 5x upper limit of normal

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2012-04-23 (Actual); Primary Completion 2014-06-13 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (55):
- United States (14):
  - Tucson, Arizona
  - Sacramento, California
  - San Diego, California
  - Jacksonville, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Syracuse, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Richmond, Virginia
- Vienna, Austria
- Bruges, Belgium
- London, Ontario, Canada
- Colombia (2):
  - Medellín, Antioquia
  - Baranquilla, Atlántico
- Aarhus N, Denmark
- France (4):
  - Bron
  - Marseille
  - Reims
  - Rennes
- Germany (2):
  - Heidelberg, Baden-Wurttemberg
  - Bonn, North Rhine-Westphalia
- Ramat Gan, Israel
- Italy (4):
  - Napoli, Campania
  - Rome, Lazio
  - Milan, Lombardy
  - Turin, Piedmont
- Japan (6):
  - Nagoya, Aichi-ken
  - Nishinomiya, Hyōgo
  - Kashihara, Nara
  - Shinjuku-ku, Tokyo
  - Suginami, Tokyo
  - Hiroshima
- Netherlands (4):
  - Amsterdam
  - Groningen
  - Maastricht
  - The Hague
- Oslo, Norway
- Wroclaw, Poland
- Timișoara, Romania
- Singapore, Singapore
- South Korea (3):
  - Busan, Busan Gwang''yeogsi
  - Daejeon
  - Seoul
- Taiwan (2):
  - Changhua
  - Taipei
- Turkey (Türkiye) (2):
  - Ankara
  - Izmir
- United Kingdom (3):
  - Newcastle upon Tyne, Vale of Glamorgan, the
  - London
  - Sheffield

REFERENCES:
- [Background] Baumann A, Piel I, Hucke F, Sandmann S, Hetzel T, Schwarz T. Pharmacokinetics, excretion, distribution, and metabolism of 60-kDa polyethylene glycol used in BAY 94-9027 in rats and its value for human prediction. Eur J Pharm Sci. 2019 Mar 15;130:11-20. doi: 10.1016/j.ejps.2019.01.015. Epub 2019 Jan 14. PMID 30654111
- [Background] Lalezari S, Reding MT, Pabinger I, Holme PA, Negrier C, Chalasani P, Shin HJ, Wang M, Tseneklidou-Stoeter D, Maas Enriquez M. BAY 94-9027 prophylaxis is efficacious and well tolerated for up to >5 years with extended dosing intervals: PROTECT VIII extension interim results. Haemophilia. 2019 Nov;25(6):1011-1019. doi: 10.1111/hae.13853. Epub 2019 Oct 17. PMID 31621991
- [Background] Reding MT, Ng HJ, Poulsen LH, Eyster ME, Pabinger I, Shin HJ, Walsch R, Lederman M, Wang M, Hardtke M, Michaels LA. Safety and efficacy of BAY 94-9027, a prolonged-half-life factor VIII. J Thromb Haemost. 2017 Mar;15(3):411-419. doi: 10.1111/jth.13597. Epub 2017 Feb 22. PMID 27992112
- [Result] Reding MT, Pabinger I, Holme PA, Maas Enriquez M, Mancuso ME, Lalezari S, Miesbach W, Di Minno G, Klamroth R, Hermans C. Efficacy and safety of damoctocog alfa pegol prophylaxis in patients ⩾40 years with severe haemophilia A and comorbidities: post hoc analysis from the PROTECT VIII study. Ther Adv Hematol. 2023 Apr 22;14:20406207231166779. doi: 10.1177/20406207231166779. eCollection 2023. PMID 37113811
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 3 parts: Part A (main study [36-week treatment period] and an optional extension [at least 100 total exposure days]) and Part B for major surgeries (up to 3 weeks).
Pre-assignment Details: Of 149 participants screened in Part A, 134 were treated, reasons for non-inclusion were screen failure, consent withdrawal, and non-adherence to protocol visit windows. Participants selected either on-demand or prophylaxis treatment at start of study according to their preference. Randomization to prophylaxis arms occurred after week 10.
Groups:
- BAY94-9027 On-demand Treatment, Part A: Participants received on-demand treatment with BAY94-9027 as an intravenous (IV) infusion at a dose as indicated based upon location and severity of bleeds (a maximum of 60 international units per kilogram [IU/kg]). Participants entering extension either continued their on-demand treatment or switched to one of the prophylaxis regimens.
- BAY94-9027 Prophylaxis Treatment, Part A: All participants started BAY94-9027 IV infusion, with 2x/week at a dose of 25 IU/kg for 10 weeks. Thereafter, participants with less than 2 spontaneous joint and/or muscle bleeds were randomized 1:1 to either every 5 or every 7 days dosing regimen. High bleeders continued 2x/week infusion (2x/week 'failed'). Participants qualified to be randomized but enrolled after randomized arms were filled, remained on 2x/week treatment (2x/week 'forced' group). Participants entering extension either continued their prophylaxis regimen or switched to one of the other prophylaxis regimens.
- BAY949027 Treatment in Major Surgery, Part B: Participants who underwent major surgery received study drug during their hospital stay up to 3 weeks post surgery. Participants were treated according to the type of procedure, using tailored doses (a maximum of 60 IU/kg/infusion) expected to maintain acceptable therapeutic level of FVIII activity.
Period: Part A_Main Trial
Arm/Group | BAY94-9027 On-demand Treatment, Part A | BAY94-9027 Prophylaxis Treatment, Part A | BAY949027 Treatment in Major Surgery, Part B
Started (Received Treatment) | 20 | 114 | 0 (Participants in Part B were not counted for Part A)
Completed | 18 | 108 | 0
Not Completed | 2 | 6 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 0
Not completed — Non-adherence to the protocol | 1 | 0 | 0
Period: Part A_Extension
Arm/Group | BAY94-9027 On-demand Treatment, Part A | BAY94-9027 Prophylaxis Treatment, Part A | BAY949027 Treatment in Major Surgery, Part B
Started | 14 (Not all participants from main trial entered extension or remained in the same arm.) | 107 (Not all participants from main trial entered extension or remained in the same arm.) | 0 (Participants in Part B were not counted for part A)
Completed | 14 | 95 | 0
Not Completed | 0 | 12 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other Reason | 0 | 1 | 0
Not completed — Completed Japan only | 0 | 5 | 0
Period: Part B
Arm/Group | BAY94-9027 On-demand Treatment, Part A | BAY94-9027 Prophylaxis Treatment, Part A | BAY949027 Treatment in Major Surgery, Part B
Started (Treated in Part B) | 0 (Time in Part A for 8 participants coming from Part A was not counted in part B.) | 0 (Time in Part A for 8 participants coming from Part A was not counted in part B.) | 19 (11 participants were enrolled in Part B only, 8 participants switched from Part A to Part B.)
Completed | 0 | 0 | 17
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other reason | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- BAY94-9027 On-demand Treatment, Main Trial: Participants received on-demand treatment with BAY94-9027 as an intravenous (IV)infusion at a dose as indicated based upon location and severity of bleeds (a maximum of 60 international units per kilogram [IU/kg]).
- BAY94-9027 Prophylaxis Treatment, 2x/Week Dropped, Main Trial: 4 participants dropped out during week 0-10
- BAY94-9027 Prophylaxis Treatment, 2x/Week Failed, Main Trial: All participants started BAY94-9027 IV infusion with 2x/week at a dose of 25 IU/kg for 10 weeks. High bleeders (with 2 or more muscle or joint bleeds in the first 10 weeks) continued 2x/week infusion (2x/week 'failed') at a dose of 30 to 40 IU/kg.
- BAY94-9027 Prophylaxis Treatment, 2x/Week Forced, Main Trial: All participants started BAY94-9027 IV infusion with 2x/week at a dose of 25 IU/kg for 10 weeks. Participants with < 2 spontaneous joint and/or muscle bleeds were randomized 1:1 to either every 5 or every 7 days dosing regimen. Participants enrolled after randomization arms were filled continued 2x/week treatment at a dose of 30-40 IU/kg (2x/week 'forced').
- BAY94-9027 Prophylaxis Treatment, Every 5 Days, Main Trial: All participants started BAY94-9027 IV infusion with 2x/week at a dose of 25 IU/kg for 10 weeks. Participants with < 2 spontaneous joint and/or muscle bleeds were randomized 1:1 to either every 5 or every 7 days dosing regimen, participants randomized to the every 5 days treatment arm were to begin treatment with 45 IU/kg every 5 days with the option to increase dose up to 60 IU/kg/infusion.
- BAY94-9027 Prophylaxis Treatment, Every 7 Days, Main Trial: All participants started BAY94-9027 IV infusion with 2x/week at a dose of 25 IU/kg for 10 weeks. Participants <2 spontaneous joint and/or muscle bleeds were randomized 1:1 to either every 5 or every 7 days dosing regimen, participants randomized to the every 7 days treatment arm were to administer a dose of 60 IU/kg (maximum 6000 IU) every 7 days.
- BAY94-9027 Treatment in Major Surgery, Part B Only: Participants treated in Part B only were included. Participants treated in Part A and continued in Part B were excluded. Participants who underwent major surgery received study drug during their hospital stay and up until hospital discharge or 3 weeks post-surgery, whichever came first. Participants were treated according to the type of procedure, using tailored doses (a maximum of 60 IU/kg) expected to maintain acceptable therapeutic level of FVIII activity.
- Total: Total of all reporting groups
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Dropped, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Failed, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Forced, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 5 Days, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 7 Days, Main Trial | BAY94-9027 Treatment in Major Surgery, Part B Only | Total
Number analyzed (Participants) | 20 | 4 | 13 | 11 | 43 | 43 | 11 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (13.5) | 27.3 (14.2) | 31.4 (11.6) | 33.1 (11.0) | 33.7 (13.0) | 37.0 (13.5) | 37.9 (13.7) | 36.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 20 | 4 | 13 | 11 | 43 | 43 | 11 | 145

OUTCOME MEASURES:

1. Primary Outcome: Annualized Number of Total Bleeds in On-demand Treatment Arm (Weeks 0 -36) and in Each Prophylaxis Arm (Weeks 10 - 36, Excluding Rescue Bleeds) - Part A, Main Trial
Description: Annualized number of total bleeds was defined as the annualized sum of spontaneous bleeds and trauma bleeds. A participant who had the one-time increase in dose frequency was regarded as rescued. A rescue bleed was a bleed that occured after the dose frequency was increased. Rescue bleeds and periods were not considered for the annualized bleeding rate (ABR).
Time Frame: On-demand: Weeks 0 -36 and Prophylaxis: Weeks 10 - 36 during Part A
Population: Intent to treat (ITT) population part A week 10-36, 4 participants dropped out during week 0-10.
Measure: Median (Inter-Quartile Range); unit: bleeds
Groups:
- BAY94-9027 Prophylaxis Treatment Total, Main Trial: All participants receiving an schedule of prophylaxis treatment, all prophylaxis arms combined.
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Failed, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Forced, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 5 Days, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 7 Days, Main Trial | BAY94-9027 Prophylaxis Treatment Total, Main Trial
Number analyzed (Participants) | 20 | 13 | 11 | 43 | 43 | 110
bleeds | 23.42 [17.84 to 37.25] | 4.11 [2.01 to 10.56] | 1.93 [0.00 to 5.24] | 1.93 [0.00 to 4.23] | 3.85 [0.00 to 6.47] | 2.09 [0.00 to 6.05]

2. Secondary Outcome: Annualized Number of Joint Bleeds, Trauma, Spontaneous Bleeds in On-demand Treatment Arm (Weeks 0 -36) and in Each Prophylaxis Arm (Weeks 10 - 36, Excluding Rescue Bleeds) - Part A
Description: A participant who had the one-time increase in dose frequency was regarded as rescued. A rescue bleed was a bleed that occured after the dose frequency was increased. Rescue bleeds and periods were not considered for the ABR.
Time Frame: On-demand: Weeks 0 -36 and Prophylaxis: Weeks 10 - 36 during Part A
Population: ITT population part A week 10-36, 4 participants dropped out during week 0-10.
Measure: Median (Inter-Quartile Range); unit: bleeds
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Failed, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Forced, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 5 Days, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 7 Days, Main Trial | BAY94-9027 Prophylaxis Treatment Total, Main Trial
Number analyzed (Participants) | 20 | 13 | 11 | 43 | 43 | 110
bleeds
  Joint Bleeds | 16.34 [11.61 to 30.30] | 4.01 [1.98 to 8.03] | 1.93 [0.00 to 5.24] | 1.86 [0.00 to 3.99] | 1.92 [0.00 to 6.26] | 1.93 [0.00 to 5.24]
  Trauma Bleeds | 9.09 [3.08 to 15.53] | 1.98 [0.00 to 5.80] | 0.00 [0.00 to 1.93] | 0.00 [0.00 to 2.09] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 1.98]
  Spontaneous Bleeds | 14.29 [7.26 to 22.71] | 3.87 [0.00 to 4.11] | 0.00 [0.00 to 1.93] | 0.00 [0.00 to 3.99] | 1.93 [0.00 to 6.33] | 0.00 [0.00 to 4.17]

3. Secondary Outcome: Annualized Number of Total Bleeds in On-demand Treatment Arm and in Each Prophylaxis Arm, Part A, Extension
Description: Annualized number of total bleeds was defined as the annualized sum of spontaneous bleeds and trauma bleeds.
Time Frame: at least 100 total exposure days acquired, median time 3.9 years up to 7 years maximum
Population: ITT extension population. Participants in each regimen stayed on this regimen without switch. Participants who switched regimen were analyzed in the variable frequency arm.
Measure: Median (Inter-Quartile Range); unit: bleeds
Groups:
- BAY94-9027 On-demand Treatment, Extension: On-demand participants entering the Part A extension either continued their on-demand treatment or switched to one of the prophylaxis regimens.
- BAY94-9027 Prophylaxis Treatment, 2x/Week, Extension; BAY94-9027 Prophylaxis Treatment, Every 5 Days, Extension; BAY94-9027 Prophylaxis Treatment, Every 7 Days, Extension: Prophylaxis participants entering the Part A extension were either to continue their prophylaxis regimen as it was at the conclusion of the main trial, or had the option of switching to one of the other prophylaxis regimens.
- BAY94-9027 Prophylaxis Treatment, Variable, Extension: Participants changed their treatment regimens at least once after 1st week in extension.
Arm/Group | BAY94-9027 On-demand Treatment, Extension | BAY94-9027 Prophylaxis Treatment, 2x/Week, Extension | BAY94-9027 Prophylaxis Treatment, Every 5 Days, Extension | BAY94-9027 Prophylaxis Treatment, Every 7 Days, Extension | BAY94-9027 Prophylaxis Treatment, Variable, Extension
Number analyzed (Participants) | 14 | 23 | 33 | 23 | 28
bleeds | 34.09 [20.33 to 36.63] | 1.57 [0.79 to 3.61] | 1.17 [0.00 to 4.57] | 0.65 [0.00 to 1.68] | 3.10 [1.13 to 5.86]

4. Secondary Outcome: Number of Participants Developed Human Coagulation Factor VIII (FVIII) Inhibitor - Part A
Description: FVIII inhibitor testing was done according to the Nijmegen modified Bethesda assay. A positive inhibitor test was defined with a threshold of ≥0.6 Bethesda unit (BU) at the central laboratory.
Time Frame: Weeks 0 to 36 during Part A
Population: Part A safety population (N=134) included all participants who received at least 1 dose of study drug during Part A of the study.
Measure: Count of Participants; unit: Participants
Groups:
- BAY94-9027 Prophylaxis Treatment, Week 0-36, Main Trial: All participants in the prophylaxis arms started BAY94-9027 IV infusion, with 2x/week at a dose of 25 IU/kg for 10 weeks. Thereafter, participants with less than 2 spontaneous joint and/or muscle bleeds were randomized 1:1 to either every 5 or every 7 days dosing regimen. High bleeders continued 2x/week infusion (2x/week 'failed'). Participants qualified to be randomized, but enrolled after randomized arms were filled, remained on 2x/week treatment (2x/week 'forced' group).
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, Week 0-36, Main Trial
Number analyzed (Participants) | 20 | 114
Participants | 0 | 0

5. Secondary Outcome: Number of Bleeds Requiring 1, 2 or >= 3 Infusions to Control the Bleed - Part A
Description: Number of bleeds requiring 1, 2 or >= 3 infusions to control the bleeding
Time Frame: Weeks 0 to 36
Population: Part A ITT population, analysis population includes participants who presented >=1 bleeding event.
Measure: Number; unit: bleeds
Units Other Than Participants: bleeds
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, Week 0-36, Main Trial
Number analyzed (Participants) | 20 | 75
Number analyzed (bleeds) | 386 | 316
bleeds
  1 infusion | 307 | 262
  2 infusions | 45 | 22
  Greater than or equal to (>=) 3 infusions | 34 | 32

6. Secondary Outcome: Number of Bleeds According to Locations - Part A
Description: Bleed locations were categorised as joint, muscle, skin/mucosa, internal, others and missing.
Time Frame: Weeks 0 -36
Population: Analysis population includes participants who presented >=1 bleeding event.
Measure: Number; unit: bleeds
Units Other Than Participants: bleeds
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, Week 0-36, Main Trial
Number analyzed (Participants) | 20 | 75
Number analyzed (bleeds) | 386 | 316
bleeds
  Missing | 0 | 0
  Joint | 303 | 235
  Muscle | 54 | 59
  Skin/Mucosa | 12 | 12
  Internal | 7 | 7
  Other | 26 | 16

7. Secondary Outcome: Number of Bleeds Over Time Since Previous Prophylaxis Infusion - Part A
Time Frame: Weeks 0 to 36
Population: Analysis population includes participants who presented >=1 bleeding event.
Measure: Number; unit: bleeds
Units Other Than Participants: bleeds
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, Week 0-36, Main Trial
Number analyzed (Participants) | 20 | 75
Number analyzed (bleeds) | 386 | 316
bleeds
  <1 day | 4 | 21
  >=1 to <2 days | 19 | 62
  >=2 to <3 days | 30 | 82
  >=3 to <4 days | 30 | 69
  >=4 to <5 days | 38 | 32
  >=5 to <6 days | 42 | 36
  >=6 to <7 days | 31 | 11
  >=7 days | 192 | 3

8. Secondary Outcome: Number of Bleeds According to Participant's Assessment of Response to Treatment - Part A
Description: Response to treatment was assessed by participant as excellent, good, moderate, poor or missing during Part A of the study.
Time Frame: Weeks 0 to 36 during Part A
Population: Analysis population includes participants who presented >=1 bleeding event.
Measure: Number; unit: bleeds
Units Other Than Participants: bleeds
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, Week 0-36, Main Trial
Number analyzed (Participants) | 20 | 75
Number analyzed (bleeds) | 386 | 316
bleeds
  Excellent or Good | 252 | 256
  Excellent | 81 | 107
  Good | 171 | 149
  Moderate | 115 | 47
  Poor | 16 | 7
  Missing | 3 | 6

9. Secondary Outcome: Recombinant Human Factor VIII (rFVIII) Usage Expressed as Total Dose Per Kilogram Per Year - Part A
Description: For prophylaxis patients, the dose is related to all infusions.
Time Frame: On-demand: Weeks 0 -36 and Prophylaxis: Weeks 10 - 36 during Part A
Population: ITT population part A week 10-36, 4 participants dropped out during week 0-10.
Measure: Median (Full Range); unit: IU/kg/year
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Failed, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Forced, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 5 Days, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 7 Days, Main Trial | BAY94-9027 Prophylaxis Treatment Total, Main Trial
Number analyzed (Participants) | 20 | 13 | 11 | 43 | 43 | 110
IU/kg/year | 1518.5 [390 to 3655] | 4421.4 [3759 to 5978] | 3314.4 [2651 to 4062] | 3482.9 [2936 to 6774] | 3338.7 [2764 to 5789] | 3421.0 [2651 to 6774]

10. Secondary Outcome: Recombinant Human Factor VIII (rFVIII) Usage Expressed as Dose Per Kilogram Per Infusion - Part A
Description: For prophylaxis patients, the dose per infusion related to prophylaxis infusion.
Time Frame: On-demand: Weeks 0 -36 and Prophylaxis: Weeks 10 - 36 during Part A
Population: ITT population part A week 10-36, 4 participants dropped out during week 0-10.
Measure: Median (Full Range); unit: IU/kg/infusion
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Failed, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Forced, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 5 Days, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 7 Days, Main Trial | BAY94-9027 Prophylaxis Treatment Total, Main Trial
Number analyzed (Participants) | 20 | 13 | 11 | 43 | 43 | 110
IU/kg/infusion | 32.8 [23 to 58] | 39.2 [33 to 42] | 30.6 [29 to 41] | 45.3 [39 to 58] | 59.0 [51 to 64] | 46.9 [29 to 64]

11. Secondary Outcome: Number of Participants Requiring an Increase in Dose Frequency, or Dose Increase, During Weeks 10 to 36 - Part A
Time Frame: Weeks 10 to 36 during Part A
Population: ITT population part A week 10-36, 4 participants dropped out during week 0-10.
Measure: Count of Participants; unit: Participants
Arm/Group | BAY94-9027 Prophylaxis Treatment, 2x/Week Failed, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Forced, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 5 Days, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 7 Days, Main Trial | BAY94-9027 Prophylaxis Treatment Total, Main Trial
Number analyzed (Participants) | 13 | 11 | 43 | 43 | 110
Participants
  Dose frequency increased | 0 | 0 | 0 | 11 | 11
  Dose increased | 2 | 0 | 7 | 0 | 9

12. Secondary Outcome: Number of Surgeries According to Physician's Assessment of Adequacy of Hemostasis in Major Surgery - Part B
Description: Major surgery was defined as any surgical or invasive procedure (elective or emergent) in which the overall bleeding risk was excessive, required a general anesthetic in an individual without a bleeding disorder, penetrated or exposed a major body cavity, resulted in substantial impairment of physical or physiological functions, or required special anatomic knowledge or manipulative skill. Adequacy of hemostasis was assessed as excellent, good, moderate or poor, by the surgeon or interventionalist during Part B of the study.
Time Frame: Day of surgery
Population: 17 participants were included in the Part B ITT population.
Measure: Number; unit: surgeries
Units Other Than Participants: surgeries
Arm/Group | BAY949027 Treatment in Major Surgery, Part B
Number analyzed (Participants) | 17
Number analyzed (surgeries) | 20
surgeries
  Good | 13
  Excellent | 7
  Moderate | 0
  Poor | 0

13. Secondary Outcome: Recombinant Human Factor VIII (rFVIII) Usage Expressed as Dose Per Kilogram Per Infusion for Major Surgery - Part B
Description: Major surgery was defined as any surgical or invasive procedure (elective or emergent) in which the overall bleeding risk was excessive, required a general anesthetic in an individual without a bleeding disorder, penetrated or exposed a major body cavity, resulted in substantial impairment of physical or physiological functions, or required special anatomic knowledge or manipulative skill. Total dose per kilogram per Infusion was expressed in international units per kilogram per infusion (IU/kg/infusion).
Time Frame: Up to 3 weeks post-surgery during Part B
Population: Part B ITT population
Measure: Median (Full Range); unit: IU/kg/infusion
Units Other Than Participants: surgeries
Arm/Group | BAY949027 Treatment in Major Surgery, Part B
Number analyzed (Participants) | 17
Number analyzed (surgeries) | 20
IU/kg/infusion | 33.7 [22 to 51]

14. Secondary Outcome: Recombinant Human Factor VIII (rFVIII) Usage Expressed as Number of Infusions for Major Surgery - Part B
Description: Major surgery was defined as any surgical or invasive procedure (elective or emergent) in which the overall bleeding risk was excessive, required a general anesthetic in an individual without a bleeding disorder, penetrated or exposed a major body cavity, resulted in substantial impairment of physical or physiological functions, or required special anatomic knowledge or manipulative skill.rFVIII usage expressed as number of infusions and IU/kg per year, as well as IU/kg per event (surgery) was assessed by investigator.
Time Frame: Up to 3 weeks post-surgery during Part B
Population: Part B ITT population
Measure: Median (Full Range); unit: infusions
Units Other Than Participants: surgeries
Arm/Group | BAY949027 Treatment in Major Surgery, Part B
Number analyzed (Participants) | 17
Number analyzed (surgeries) | 20
infusions | 8.0 [3 to 39]

15. Secondary Outcome: Maximum Drug Plasma Concentration (Cmax) Following Single and Multiple Doses of BAY94-9027, Chromogenic Assay - Part A
Description: Cmax: Maximum observed drug concentration following an infusion of 60 IU/kg
Time Frame: Weeks 0 and 36: pre-infusion (0 hours), post-infusion 15, 30 minutes, 1, 3, 6, 8, 24, 48, 72, 96 hours
Population: Pharmacokinetic Analysis Set (PKS) with participants evaluable for this outcome, PKS included all participants with a valid profile of BAY94-9027 during Part A of the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: IU/dL
Groups:
- BAY94-9027 Treatment - Part A, Week 0: Part A, Week 0 included all PKS participants treated with a single (first) dose of BAY94-9027 as an IV infusion at Week 0.
- BAY94-9027 Treatment - Part A, Week 36: Part A, Week 36 group included all PKS participants treated with multiple doses (last dose paired) of BAY94-9027 as an IV infusion at Week 36. Paired data were defined as the single dose data for the sub-set of participants who also had multiple dose PK data.
Arm/Group | BAY94-9027 Treatment - Part A, Week 0 | BAY94-9027 Treatment - Part A, Week 36
Number analyzed (Participants) | 22 | 15
IU/dL | 162.8 (14.74) | 177.1 (20.98)

16. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC) Following Single and Multiple Doses of BAY94-9027, Chromogenic Assay - Part A
Description: AUC: The total area under the plasma concentration versus time curve following an infusion of 60 IU/kg .
Time Frame: Weeks 0 and 36: pre-infusion (0 hours), post-infusion 15, 30 minutes, 1, 3, 6, 8, 24, 48, 72, 96 hours
Population: PKS with participants evaluable for this outcome
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*IU/dL
Arm/Group | BAY94-9027 Treatment - Part A, Week 0 | BAY94-9027 Treatment - Part A, Week 36
Number analyzed (Participants) | 22 | 15
h*IU/dL | 3707.5 (33.77) | 4130.8 (28.8)

17. Secondary Outcome: Terminal Elimination Half Life (t1/2) Following Single and Multiple Doses of BAY94-9027, Chromogenic Assay - Part A
Description: t1/2: Terminal half-life is the time the plasma concentration during terminal phase is halved following an infusion of 60 IU/kg .
Time Frame: Weeks 0 and 36: pre-infusion (0 hours), post-infusion 15, 30 minutes, 1, 3, 6, 8, 24, 48, 72, 96 hours
Population: PKS with participants evaluable for this outcome
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | BAY94-9027 Treatment - Part A, Week 0 | BAY94-9027 Treatment - Part A, Week 36
Number analyzed (Participants) | 22 | 15
Hours | 17.1 (27.05) | 19.6 (38.48)

18. Secondary Outcome: Overall Human Coagulation Factor VIII (FVIII) Recovery Value by Chromogenic Assay - Part A
Description: Recovery was calculated by the following formula: Recovery = (post-infusion FVIII activity - pre-infusion FVIII activity ) * weight / dose (in IU). Recovery is the increase of FVIII activity after the injection normalized by dose: IU/dl per IU/kg = kg/dL
Time Frame: Weeks 0 to 36 during Part A
Population: Part A ITT population
Measure: Mean (Standard Deviation); unit: Kilogram per deciliter
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, Week 0-36, Main Trial
Number analyzed (Participants) | 20 | 112
Kilogram per deciliter | 2.67 (0.54) | 2.68 (0.55)

19. Secondary Outcome: Change From Baseline in Quality of Life by Hemophilia Specific Quality of Life Instrument or Questionnaire for Adults (Haemo-QoL-A) Overall Score at Week 36 - Part A
Description: Quality of life (QoL) was measured by the Haemo-QoL-A overall score, which ranged from 0 (the worst condition) to 100 (the best condition).
Time Frame: Week 0 (baseline) and Week 36 during Part A
Population: Part A ITT population with participants evaluable for this outcome
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, Week 0-36, Main Trial
Number analyzed (Participants) | 19 | 97
scores on a scale | -0.14 (9.70) | 2.59 (7.98)

20. Other Pre Specified Outcome: Change From Baseline in Overall Pain Severity and Interference Due to Pain at Week 36 - Part A
Description: Brief Pain Inventory (BPI) - Short Form (BPI-SF) was a 15-item, self-administered, validated tool developed to assess pain used in the study for patient reported outcomes. Scores ranged from 0 to 10 and a higher score indicates a higher level of pain/interference.
Time Frame: Week 0 (baseline) and Week 36 during Part A
Population: Analysis population includes participants evaluable in each category for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, Week 0-36, Main Trial
Number analyzed (Participants) | 20 | 112
scores on a scale
  Pain severity subscale: number analyzed (Participants) | 15 | 78
  Pain severity subscale | -0.8 (1.8) | 0.1 (1.39)
  Interference subscale: number analyzed (Participants) | 15 | 77
  Interference subscale | -0.99 (2.54) | -0.06 (1.39)

21. Other Pre Specified Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire at Week 36 - Part A
Description: The WPAI is a validated instrument to assess the effect of hemophilia on ability to work, attend classes, and perform regular daily activities in participants aged 12 and above. The WPAI also contained classroom impairment questions (CIQ). The questionnaire was self-administered and comprised of nine questions that elicited information on work, classroom, and daily activity impairment during the previous seven days. WPAI outcomes that are overall work and activity impairment, transformed to impairment percentages (range from 0 to 100), with higher numbers indicating greater impairment and less productivity.
Time Frame: Week 0 (baseline) and Week 36 during Part A
Population: Analysis population includes participants evaluable in each category for this outcome.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment Total, Main Trial
Number analyzed (Participants) | 20 | 112
scores on a scale
  Activity impairment: number analyzed (Participants) | 20 | 108
  Activity impairment | 4.74 (24.12) | -7.13 (20.00)
  Overall work impairment: number analyzed (Participants) | 12 | 62
  Overall work impairment | 4.44 (21.94) | -1.22 (21.94)

22. Other Pre Specified Outcome: Recombinant Human Factor VIII (rFVIII) Usage Expressed as Number of Infusions- Part A
Description: For prophylaxis patients, the dose is related to all infusions.
Time Frame: On-demand: Weeks 0 -36 and Prophylaxis: Weeks 10 - 36 during Part A
Population: ITT population part A week 10-36, 4 participants dropped out during week 0-10.
Measure: Median (Full Range); unit: infusions
Arm/Group | BAY94-9027 On-demand Treatment, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Failed, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Forced, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 5 Days, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 7 Days, Main Trial | BAY94-9027 Prophylaxis Treatment Total, Main Trial
Number analyzed (Participants) | 20 | 13 | 11 | 43 | 43 | 110
infusions | 29 [9 to 76] | 56.0 [52 to 71] | 55.0 [47 to 59] | 38.0 [3 to 58] | 27.0 [5 to 63] | 37.5 [3 to 71]

23. Other Pre Specified Outcome: Recombinant Human Factor VIII (rFVIII) Usage Expressed as Dose Per Kilogram With Prophylaxis Treatment - Part A
Description: For prophylaxis patients, the dose per kilogram is related to prophylaxis infusions.
Time Frame: Weeks 10 - 36 during Part A
Population: ITT population part A week 10-36, 4 participants dropped out during week 0-10.
Measure: Median (Full Range); unit: IU/kg
Arm/Group | BAY94-9027 Prophylaxis Treatment, 2x/Week Failed, Main Trial | BAY94-9027 Prophylaxis Treatment, 2x/Week Forced, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 5 Days, Main Trial | BAY94-9027 Prophylaxis Treatment, Every 7 Days, Main Trial | BAY94-9027 Prophylaxis Treatment Total, Main Trial
Number analyzed (Participants) | 13 | 11 | 43 | 43 | 110
IU/kg | 1986.9 [1733 to 2236] | 1669.1 [1430 to 1947] | 1704.3 [139 to 2049] | 1530.2 [122 to 1788] | 1644.9 [122 to 2236]

24. Other Pre Specified Outcome: Number of Minor Surgeries According to Physician's Assessment of Adequacy of Hemostasis - Part A
Description: Minor surgery was defined as any surgical procedure that did not meet the definition of major, and included simple dental extractions, incision and drainage of abscesses, or simple excisions.
Time Frame: Weeks 0 to 36 during Part A
Population: Part A ITT population
Measure: Number; unit: minor surgeries
Units Other Than Participants: minor surgeries
Groups:
- BAY94-9027 Treatment - Part A: This group included both on-demand and prophylaxis arms in Part A.
Arm/Group | BAY94-9027 Treatment - Part A
Number analyzed (Participants) | 10
Number analyzed (minor surgeries) | 17
minor surgeries
  Excellent | 9
  Good | 6
  Missing | 2

25. Other Pre Specified Outcome: Number of Surgeries According to Physician's Assessment of Response to Hemostasis, Post-surgery - Part B Main Trial
Description: Response to treatment during surgery was assessed by investigator/surgeon as excellent, good, moderate, poor or missing during Part B of the study.
Time Frame: Up to 3 weeks post-surgery during Part B
Population: Part B ITT population
Measure: Number; unit: surgeries
Units Other Than Participants: surgeries
Arm/Group | BAY949027 Treatment in Major Surgery, Part B
Number analyzed (Participants) | 14
Number analyzed (surgeries) | 17
surgeries
  Excellent | 8
  Good | 5
  Moderate | 3
  Missing | 1

26. Other Pre Specified Outcome: Number of Participants With Change/Drop in Hemoglobin/Hematocrit Laboratory Assessments - Part B
Description: Hematocrit is defined as the volume percentage (%) of red blood cells in blood.
Time Frame: Up to 3 weeks post-surgery during Part B
Population: Part B Safety population (N=17) included all participants who received at least 1 dose of study drug during Part B of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | BAY949027 Treatment in Major Surgery, Part B
Number analyzed (Participants) | 17
Participants
  Hematocrit | 6
  Hemoglobin | 2

27. Other Pre Specified Outcome: Maximum Blood Loss During Major Surgery - Part B
Description: Major surgery was defined as any surgical or invasive procedure (elective or emergent) in which the overall bleeding risk was excessive, required a general anesthetic in an individual without a bleeding disorder, penetrated or exposed a major body cavity, resulted in substantial impairment of physical or physiological functions, or required special anatomic knowledge or manipulative skill.
Time Frame: day of surgery
Population: Part B ITT population with participants treated for major surgery
Measure: Number; unit: milliliter
Units Other Than Participants: surgeries
Arm/Group | BAY949027 Treatment in Major Surgery, Part B
Number analyzed (Participants) | 17
Number analyzed (surgeries) | 20
milliliter | 1000

28. Other Pre Specified Outcome: Number of Participants Who Took Anti-fibrinolytic Medications During Major Surgery - Part B
Description: as for outcome 27
Time Frame: Up to 3 weeks post-surgery during Part B
Population: Part B ITT population with participants treated for major surgery
Measure: Count of Participants; unit: Participants
Arm/Group | BAY949027 Treatment in Major Surgery, Part B
Number analyzed (Participants) | 17
Participants | 8

29. Other Pre Specified Outcome: Volume of Blood Transfused in Major Surgery - Part B
Description: as for outcome 27
Time Frame: Up to 3 weeks post-surgery during Part B
Population: Part B ITT population who had blood transfusions during major surgery
Measure: Median (Full Range); unit: milliliter
Units Other Than Participants: surgeries
Arm/Group | BAY949027 Treatment in Major Surgery, Part B
Number analyzed (Participants) | 4
Number analyzed (surgeries) | 5
milliliter | 865 [600 to 1380]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected after the first dose of study drug and up to 7 days after the last dose over a period of approximately 5 years.
Groups:
- BAY94-9027 Treatment, Part A, Main Trial: Subjects entering Part A main trial were treated with BAY 94-9027 for either on-demand or prophylactic treatment.
- BAY94-9027 Treatment, Part A, Extension: Subjects in Part A extension either continued their regimen from main trial or switched to one of the other regimens at any time.
- BAY94-9027 Treatment in Major Surgery, Part B: Subjects, either Part B subjects only or subjects from Part A/Part A Extension, who underwent major surgery received study drug during their hospital stay up to 3 weeks post-surgery. Subjects were treated according to the type of procedure, using tailored doses (a maximum of 60 IU/kg/infusion) expected to maintain acceptable therapeutic level of FVIII activity.
Arm/Group | BAY94-9027 Treatment, Part A, Main Trial | BAY94-9027 Treatment, Part A, Extension | BAY94-9027 Treatment in Major Surgery, Part B
All-Cause Mortality (participants affected / at risk) | 0/134 | 0/121 | 0/22
Serious Adverse Events (participants affected / at risk) | 13/134 | 36/121 | 2/22
Other Adverse Events (participants affected / at risk) | 67/134 | 74/121 | 16/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY94-9027 Treatment, Part A, Main Trial (N=134) | BAY94-9027 Treatment, Part A, Extension (N=121) | BAY94-9027 Treatment in Major Surgery, Part B (N=22)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasal vestibulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anti factor VIII antibody positive (Investigations) | 0 (0) | 0 (0) | 2 (2)
Colonoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Renal stone removal (Surgical and medical procedures) | 0 (0) | 1 (2) | 0 (0)
Ureteral stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY94-9027 Treatment, Part A, Main Trial (N=134) | BAY94-9027 Treatment, Part A, Extension (N=121) | BAY94-9027 Treatment in Major Surgery, Part B (N=22)
Nausea (Gastrointestinal disorders) | 5 (6) | 5 (7) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 10 (13) | 3 (3)
Influenza (Infections and infestations) | 5 (9) | 8 (12) | 0 (0)
Nasopharyngitis (Infections and infestations) | 24 (34) | 25 (55) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 7 (9) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 12 (14) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) | 8 (8) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 7 (8) | 9 (10)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (13) | 26 (40) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 14 (17) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (10) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (12) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (11) | 0 (0)
Headache (Nervous system disorders) | 16 (28) | 14 (21) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 9 (11) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 6 (6) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Some registered "Secondary outcome measure" were re-classified as "Other Pre-specified" in line with protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less